CLINICAL TRIAL: NCT01935284
Title: Post-Market Study Evaluating Analyzer Readings of Multiple Arterial Blood Gas Syringes
Brief Title: Evaluation of Blood Gas Syringes
Acronym: Analyze ABS
Status: Completed | Type: Observational
Sponsor: Smiths Medical, ASD, Inc. (Industry)
Collaborators: Bionostics (Unknown)
Responsible Party: Sponsor
Other Study IDs: Analyze ABS
Record Dates: First submitted 2013-06-26; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Blood Gas Analyte Values

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers

SUMMARY:
To assess the interchangeability and agreement between measurements from three blood gas syringes for the collection of blood for the analysis of multiple analytes as measured by differing manufacturers' multi-parameter analyzers.

DETAILED DESCRIPTION:
This is a prospective, randomized, post-market study using fresh blood for analysis that is obtained from healthy subject volunteers. Trained phlebotomists will collect blood samples from subjects after confirmation of eligibility criteria. Blood samples will be drawn to fill all study syringe types in a randomized order. Each syringe type will be drawn per subject to analyze each of the available blood parameters in duplicate using three different multi-parameter analyzers. The analytes tested will vary per analyzer capabilities. All blood draws and analyte testing will be performed at an independent laboratory. The study is to confirm that all of the syringes tested provide consistent readings when analyzed using the most common multi-parameter analyzers used in hospital laboratories.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Willing and able to independently sign an English Informed Consent
3. Have adequate veins for sampling blood from both right and left upper extremities

Exclusion Criteria:

1. Currently taking anti-coagulation medication
2. Have a known bloodborne disease or bleeding tendency
3. Have a known fear or adverse reaction to needles or blood
4. Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Differences in analyte values obtained from three different blood gas syringes for each analyzer tested | Blood analysis within 30 minutes of draw
  For each of the analytes that are tested, the analyte values from each of the three (3) syringe types tested will be compared for each of the three (3) multi-parameter analyzers. Average values for each analyte per patient, syringe and analyzer will be used for the comparison of syringes for each analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cifaldi, BS, RRT, Principal Investigator — Smiths Medical
Locations (1):
- Bionostics, Devens, Massachusetts, United States